CLINICAL TRIAL: NCT01942889
Title: Antioxidants Supplementation Associated With Pulmonary Rehabilitation is it Effective on Muscle Dysfunction and Signaling Pathways Involved in the Myopathy of COPD?
Brief Title: Antioxidants and Pulmonary Rehabilitation in COPD Patients
Acronym: AREB-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: 5 Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 8710
Record Dates: First submitted 2013-08-14; First posted 2013-09-16 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD
Keywords: COPD; exercise training; pulmonary rehabilitation; antioxidant; muscle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antioxidant Supplementation (Active Comparator): Vitamin antioxidant and trace elements combination that won't exceed the maximal nutritional dose recommended in France (Vit E, vit C, Selenomethionine, Zinc gluconate).
  Interventions: Dietary Supplement: Antioxidant Supplementation associated to Comprehensive respiratory Rehabilitation Program
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Antioxidant Supplementation associated to Comprehensive respiratory Rehabilitation Program

INTERVENTIONS:
Dietary Supplement: Antioxidant Supplementation associated to Comprehensive respiratory Rehabilitation Program — Vit E, Vit C, Selenomethionine, Zinc gluconate

SUMMARY:
On the basis of published data and investigators results indicating that systemic redox in balance may contribute to the peripheral muscle dysfunction in COPD patients, the investigators propose a study testing the effects of antioxidants and exercise training in COPD patients. The results may have major implication in the improvement of pulmonary rehabilitation benefits

DETAILED DESCRIPTION:
COPD will constitute the third cause of mortality in 2012. This chronic respiratory disease is characterized by peripheral dysfunction of skeletal muscle which is associated with major clinical outcomes (prognostics, symptoms, and health related quality of life). Muscle and systemic oxidative stress has been incriminated in this peripheral muscle dysfunction.Exercise training constitute the main validated therapeutic intervention leading to significant muscle function and clinical improvement.Our preliminary results have shown that COPD patients experiment dietary and enzymatic antioxidants defects.Yet, generic antioxidant supplementation has not shown significant muscle function improvement.Therefore, we aim to test the effects of an antioxidant supplementation targeted on the antioxidant defects associated with exercise training on the peripheral muscle function, exercise tolerance and health quality of life in COPD patients.At the cellular level, this muscle dysfunction is related with a fiber atrophy and a metabolic switch (reduce proportion of oxidative fiber).This study will compare the effects of an antioxidant supplementation on the peripheral muscle function and skeletal muscle cellular properties in association with exercise training during a pulmonary rehabilitation course.Volunteers will be randomised in 2 groups: - 1 group treated with the antioxidant supplementation ( 28 days)- 1 group treated with the placeboIntervention will be allocated by chance and a double blind manner. Antioxidant supplementation will associate vitamins and trace elements that won't exceed the maximal nutritional dose recommended.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients, 40 years to 78 years, last exacerbation dating at least 4 weeks

Exclusion Criteria:

* unstabilized primary pathologies (cardiovascular, renal, metabolic, psychiatric)
* nutritional supplementation in the 4 weeks preceding the study (antioxidant, vitamins…)

Ages: 40 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
quadriceps endurance time.Time frame: at the start and the end of the study | up to day 37
  sitting on a bench, starting from a 90° knee flexion of the dominant leg, the subjects should perform knee extensions (6 movements per minute) with a workload to 30% of the isometric maximal voluntary contraction until exhaustion. The duration of the test (in seconds) characterizes the quadriceps endurance.

SECONDARY OUTCOMES:
muscle and /or serum oxidative stress level | up to day 37
  Description: oxidative stress will be evaluated by measuring lipid peroxidation and oxidized proteins.GSH/ GSSG ratio and enzymatic/non enzymatic antioxidants
Isometric maximal voluntary contraction of the quadriceps | up to day 37
  sitting on a bench with a force sensor connected to a data acquisition and analysis system signal, subjects should reproduce three trials spaced 1 minute, by an extension movement of the knee joint against a stationary load, maximum way, keeping the arms crossed over the chest and leaning against the back in order to limit the involvement of other muscles. The most elevated of the three tests repeatable value close to 10% characterizes the maximum strength of subjects.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique du souffle la vallonie, Lodève
  - University Hospital of Montpellier, Montpellier

REFERENCES:
- [Derived] Gouzi F, Maury J, Heraud N, Molinari N, Bertet H, Ayoub B, Blaquiere M, Bughin F, De Rigal P, Poulain M, Pincemail J, Cristol JP, Laoudj-Chenivesse D, Mercier J, Prefaut C, Pomies P, Hayot M. Additional Effects of Nutritional Antioxidant Supplementation on Peripheral Muscle during Pulmonary Rehabilitation in COPD Patients: A Randomized Controlled Trial. Oxid Med Cell Longev. 2019 Apr 17;2019:5496346. doi: 10.1155/2019/5496346. eCollection 2019. PMID 31178967